CLINICAL TRIAL: NCT06333067
Title: Safety and Efficacy of SofWave Treatment to Lift Facial Lax Skin and Improve Facial Wrinkles Using Precise and Lift Applicators
Brief Title: Treatment to Lift Facial Lax Skin and Improve Facial Wrinkles Using Precise and Lift Applicators
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sofwave Medical LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sofwave21
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Lax Skin
Keywords: neck zones.; submental; Facial; Skin laxity
MeSH Terms: conditions — Cutis Laxa; Facies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- lax tissue (Experimental)
  Interventions: Device: Sofwave

INTERVENTIONS:
Device: Sofwave — The Sofwave System, comprised of an applicator and a console, generates high intensity, non-focused ultrasonic energy which can be delivered percutaneously to tissues.
  Other Names: SUPERB

SUMMARY:
Open-label, non-randomized single-arm prospective, multi-center, self-controlled clinical study with masked evaluation.

DETAILED DESCRIPTION:
Eligible patients will receive 1-2 face and/or neck and/or submental treatments (per PI discretion, 2-12 weeks apart) using the SofWave system with the Lift or/and Precise applicators.

Treatment may be administered after the enrollment and screening at the first visit, or it may occur at a later date following the enrollment and screening activities based on site scheduling availabilities.

All patients will return to the clinic for one follow-up visit at 3 months ± 2 weeks post last treatment (FU1).

Methodology described in the protocol to evaluate efficacy and safety of treatments will be carried out at each visit at the clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female and male subjects between the ages 35-80.
2. Non-Smoker.
3. Fitzpatrick skin type I-VI.
4. Desire to lift facial lax skin, neck and/or submental and/or to lift the eyebrow area and/or improve facial wrinkles appearance.
5. Able and willing to comply with all visits, treatments and evaluation schedules and requirements.
6. Able to understand and provide written Informed Consent.
7. Women of child-bearing age are required to be using a reliable method of birth control at least 3 months prior to study enrollment.
8. Subject agrees not to undergo any other facial cosmetic treatment for a period of 3 months following last SofWave treatment.
9. Stable weight over the last 12 weeks and throughout the duration of the study.

Exclusion Criteria:

* 1. Pregnant or planning to become pregnant, having given birth less than 3 months ago, and/or breast feeding.

  2. Presence of any active systemic or local infections.

  3. Presence of active local skin disease that may alter wound healing.

  4. Severe solar elastosis.

  5. Currently a smoker or has a history of heavy smoking (25 cigarettes per day or more) in the past 10 years.

  6. History of chronic drug or alcohol abuse.

  7. Excessive subcutaneous fat on the cheeks.

  8. Significant scarring in the area to be treated.

  9. Severe or cystic facial acne, and/or Accutane use during past 6 months.

  10. Presence of a metal stent or implant in the facial area (dental implants and/or braces are not excluded).

  11. Inability to understand the protocol or to provide a signed informed consent.

  12. History of cosmetic treatments in the facial area to be treated, including facial skin-tightening procedure within the past 6 months; injectable (Botox or fillers) of any type within the past 6 months; ablative or non-ablative resurfacing/rejuvenation laser treatment or light treatment within the past 6 months, dermabrasion or deep facial peels within the past 12 months; facelift, blepharoplasty, or brow lift (including contour threads) within the past 12 months.

  13. Taking Isotretinoin or other oral retinoid within the past 6 months; taking anti-platelet or anti-coagulant within the past 2 weeks.

  14. As per the investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-10-11 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in the appearance of lax skin | 3 months post treatment follow-up visit
  Rate of improvement in the appearance of lax skin on the submental, neck zones and facial wrinkles following Sofwave treatments based on Global Aesthetic Improvement Scale, as evaluated by independent masked reviewers.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Costal Skin & Eye Institute, La Mesa, California
  - Skin Wellness Dermatology Associates, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided